CLINICAL TRIAL: NCT06319417
Title: Assessing the Impact of Hydroxytyrosol Caramel Treatment on the Cardiometabolic Health of Patients at Cardiovascular Risk Disease
Brief Title: Hydroxytyrosol Caramel Treatment on Cardiovascular Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, LUIS TEJADA PORTERO, Researcher, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HT-UCAM
Record Dates: First submitted 2024-03-05; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Pathology
Keywords: hydroxytyrosol; cardiovascular risk; crossover; randomized
MeSH Terms: interventions — 3,4-dihydroxyphenylethanol

STUDY DESIGN:
Intervention Model Description: 28 days of treatment: one group with HT treatment and the other with placebo treatment.
  2-weeks washout period. The treatment will be switched between groups for another 28 days: those who initially consumed HT will the switch to the placebo treatment, and vice versa.
Who Masked: Participant, Care Provider
Masking Description: Nor participant and care provider knew the treatment given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HT treatment (Experimental): Every caramel contained 15 mg of HT, cyclodextrins and xylitol. Patients consumed 4 caramels/day, totalling 60 mg of HT/day.
  Interventions: Dietary Supplement: HT treatment
- Placebo treatment (Placebo Comparator): Every caramel contained cyclodextrins and xylitol. Patients consumed 4 caramels/day.
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: HT treatment — Total consumption of 60 mg/day of HT
  Other Names: Hydroxytyrosol
  Arms: HT treatment
Dietary Supplement: Placebo treatment — Consumption of placebo treatment of 4 caramels/day
  Other Names: Placebo
  Arms: Placebo treatment

SUMMARY:
The goal of this double-blind crossover randomized clinical trial is to evaluate the impact of a phenolic natural compound called hydroxytyrosol (HT) on patients at cardiovascular risk (CVR). The main questions it aims to answer are:

* Evaluating the effect of HT caramels on CVR biomarkers.
* Assessing the impact of HT caramels on cellular phenotype.

Participants will take 4 caramels/day, each containing 15 mg of HT, consuming a daily intake of 60 mg for 28 days. One group will begin with HT caramel consumption for 28 days, while the other group will start with a placebo treatment. Following a 2-week washout period, the treatments will be switched between the groups. Those who initially consumed HT will then switch to the placebo treatment, and vice-versa, each for a duration of 28 days.

DETAILED DESCRIPTION:
A 10-week randomized, crossover, double-blind controlled clinical trial was conducted between April 2022 and March 2023 in the Catholic University of Murcia Randomization divided the participants in two groups, depending on whether they started consuming the caramels supplemented with HT, or the group that started consuming the placebo caramels.

The patients totally consumed 60 mg of HT per day distributed into 4 caramels/day with 15 mg of HT per caramel. The caramels in treatment group contained encapsulated HT in cyclodextrins, xylitol sweetened. On the other hand, the caramels in placebo group contained cyclodextrins and they were xylitol sweetened too. Patients were segregated into 2 groups: the ones who started as HT-group and the ones who started as C-group.

HT-group consumed HT caramels for 28 days, while C-group consumed placebo caramels followed by a 2-week washout period. Suddenly, groups were switched for 28 days, the ones who started as HT-group became C-group and vice-versa. The patients completely performed 4 visits during the study. In every appointment, they had blood and faeces extraction with body composition measurement. In addition, a Food Frequency Questionnaire (FFQ) based on Mediterranean Diet Serving Score (MDSS) was given to the patients in order to assess diet variability during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Elevated cholesterol level: >200 mg/dL
* Elevated glucose level: >100 mg/dL

Exclusion Criteria:

* Not been under antihypertensive, antidiabetic and/or hypoglycaemic agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Change of cardiovascular biomarkers | up to 4 months
  Evaluating the effect of HT caramels on cardiovascular biomarkers in blood samples (mg/dL)
Change of cellular phenotype of platelets | up to 2 months
  Assessing the impact of HT caramels on cellular phenotype measured with flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia (UCAM), Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noguera-Navarro C, Vinten KT, Aunon-Calles D, Carazo-Diaz C, Janssens GE, Montoro-Garcia S. Multi-omic analysis and platelet function distinguish treatment responses to hydroxytyrosol in cardiovascular risk. Food Funct. 2025 Jul 14;16(14):5928-5948. doi: 10.1039/d5fo00874c. PMID 40619979

DOCUMENTS (1):
  • Informed Consent Form (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT06319417/ICF_000.pdf